CLINICAL TRIAL: NCT00356213
Title: Laparoscopic Sleeve Gastrectomy or Laparoscopic Proximal Roux-Y-gastric Bypass in the Treatment of Morbid Obesity
Brief Title: Comparison of Laparoscopic Sleeve Gastrectomy and Roux-Y-gastric Bypass in the Treatment of Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Peterli1
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Morbid Obesity
Keywords: morbid obesity; bariatric surgery; sleeve-gastrectomy; Roux-Y-gastric bypass; outcome; weight loss
MeSH Terms: conditions — Obesity, Morbid; Weight Loss | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): laparoscopic sleeve gastrectomy
  Interventions: Procedure: sleeve gastrectomy
- B (Active Comparator): laparoscopic gastric bypass
  Interventions: Procedure: Roux-Y-gastric bypass

INTERVENTIONS:
Procedure: sleeve gastrectomy — laparoscopic sleeve gastrectomy
  Other Names: bariatric operation
  Arms: A
Procedure: Roux-Y-gastric bypass — laparoscopic gastric bypass
  Other Names: bariatric operation
  Arms: B

SUMMARY:
The laparoscopic sleeve-gastrectomy (SG) compared to laparoscopic proximal Roux-Y-gastric bypass (PGB) is as successful in the treatment of morbid obesity in the majority of patients. In case of insufficient weight loss malabsorption can to be added by performing laparoscopic bilious-pancreatic diversion duodenal switch (BPD). The resection of the gastric fundus (LG) leads to changes in gastrointestinal hormones that are possibly different to bypassing the fundus (PGB).

DETAILED DESCRIPTION:
Background

Obesity is reaching epidemic proportions in the developed world. In morbidly obese patients only surgical treatment (bariatric operations) leads to a sustained weight loss and cure of comorbidities in the majority of patients. There exist a number of different operations resulting in either a restrictive effect and/or malabsorption, accompanied by a humoral effect which is caused by changes of the different gastrointestinal hormones. It is still unknown which patients needs which operation.

Working Hypothesis

The laparoscopic sleeve-gastrectomy (SG) compared to laparoscopic proximal Roux-Y-gastric bypass (PGB) is as successful in the treatment of morbid obesity in the majority of patients. In case of insufficient weight loss malabsorption can to be added by performing laparoscopic bilious-pancreatic diversion duodenal switch (BPD). The resection of the gastric fundus (LG) leads to changes in gastrointestinal hormones that are possibly different to bypassing the fundus (PGB).

Specific Aims

We plan to compare the SG and PGB in a prospective randomized study. Primary outcome measure is effectiveness in terms of weight loss, reduction in co-morbidity and quality of life, secondary outcome measures are early morbidity, duration and cost of the operation, late morbidity, re-operations (for complications, for insufficient weight loss), postoperative changes of gastrointestinal hormones.

Experimental Design/Methods

An interdisciplinary team evaluates morbidly obese patients for bariatric surgery. After informed consent eligible patients will be randomized into SG or PGB, a number of 45 per group. Preoperative examination consists of: quantification of comorbidity, eating behavior, indirect calorimetry, body composition by dual energy x-ray absorptiometry (DEXA), routine blood chemistry, gastrointestinal hormones before and after test meal, gastroscopy, manometry of the esophagus, upper GI series, abdominal ultrasound, quality of life. Perioperative investigations: operative time, fat tissue samples (omental and subcutaneous), early morbidity, gastrointestinal hormones before and after test meal, duration of hospital stay, costs; Follow-up data will be obtained every 3 months in the first year, twice in the second year and once per year thereafter: weight, reduction in comorbidities, blood tests, gastrointestinal hormones before and after test meal, DEXA and quality of life.

ELIGIBILITY:
Swiss patients with approval by health insurance

Patients from outside Switzerland: only if patients or their insurance will cover the costs

Inclusion Criteria:

* BMI>40

Exclusion Criteria:

* contraindication for bariatric surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2006-10-30 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
effectiveness in terms of weight loss, reduction in co-morbidity and quality of life | 5 years

SECONDARY OUTCOMES:
early morbidity, duration and cost of the operation, late morbidity, re-operations (for complications, for insufficient weight loss), postoperative changes of gastrointestinal hormones. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Peterli, Dr., Principal Investigator — Leitender Arzt, Allgemeinchirurgische Abteilung, St.Claraspital, CH-4016 Basel

REFERENCES:
- [Derived] Kraljevic M, Susstrunk J, Wolnerhanssen BK, Peters T, Bueter M, Gero D, Schultes B, Poljo A, Schneider R, Peterli R. Long-Term Outcomes of Laparoscopic Roux-en-Y Gastric Bypass vs Laparoscopic Sleeve Gastrectomy for Obesity: The SM-BOSS Randomized Clinical Trial. JAMA Surg. 2025 Apr 1;160(4):369-377. doi: 10.1001/jamasurg.2024.7052. PMID 39969869
- [Derived] Peterli R, Hurme S, Bueter M, Gronroos S, Helmio M, Salminen P. Standardized Assessment of Metabolic Bariatric Surgery Outcomes: Secondary Analysis of 2 Randomized Clinical Trials. JAMA Surg. 2024 Mar 1;159(3):306-314. doi: 10.1001/jamasurg.2023.6254. PMID 38055284
- [Derived] Saux P, Bauvin P, Raverdy V, Teigny J, Verkindt H, Soumphonphakdy T, Debert M, Jacobs A, Jacobs D, Monpellier V, Lee PC, Lim CH, Andersson-Assarsson JC, Carlsson L, Svensson PA, Galtier F, Dezfoulian G, Moldovanu M, Andrieux S, Couster J, Lepage M, Lembo E, Verrastro O, Robert M, Salminen P, Mingrone G, Peterli R, Cohen RV, Zerrweck C, Nocca D, Le Roux CW, Caiazzo R, Preux P, Pattou F. Development and validation of an interpretable machine learning-based calculator for predicting 5-year weight trajectories after bariatric surgery: a multinational retrospective cohort SOPHIA study. Lancet Digit Health. 2023 Oct;5(10):e692-e702. doi: 10.1016/S2589-7500(23)00135-8. Epub 2023 Aug 29. PMID 37652841
- [Derived] Peterli R, Wolnerhanssen BK, Peters T, Vetter D, Kroll D, Borbely Y, Schultes B, Beglinger C, Drewe J, Schiesser M, Nett P, Bueter M. Effect of Laparoscopic Sleeve Gastrectomy vs Laparoscopic Roux-en-Y Gastric Bypass on Weight Loss in Patients With Morbid Obesity: The SM-BOSS Randomized Clinical Trial. JAMA. 2018 Jan 16;319(3):255-265. doi: 10.1001/jama.2017.20897. PMID 29340679
- [Derived] Peterli R, Steinert RE, Woelnerhanssen B, Peters T, Christoffel-Courtin C, Gass M, Kern B, von Fluee M, Beglinger C. Metabolic and hormonal changes after laparoscopic Roux-en-Y gastric bypass and sleeve gastrectomy: a randomized, prospective trial. Obes Surg. 2012 May;22(5):740-8. doi: 10.1007/s11695-012-0622-3. PMID 22354457
- [Derived] Peterli R, Wolnerhanssen B, Peters T, Devaux N, Kern B, Christoffel-Courtin C, Drewe J, von Flue M, Beglinger C. Improvement in glucose metabolism after bariatric surgery: comparison of laparoscopic Roux-en-Y gastric bypass and laparoscopic sleeve gastrectomy: a prospective randomized trial. Ann Surg. 2009 Aug;250(2):234-41. doi: 10.1097/SLA.0b013e3181ae32e3. PMID 19638921